CLINICAL TRIAL: NCT07087431
Title: PROACT 3: Impact of Disclosing Coronary Artery Disease Polygenic Risk Score on Cardiovascular Health
Brief Title: Impact of Disclosing Coronary Artery Disease Polygenic Risk Score on Cardiovascular Health
Acronym: PROACT 3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Akl C. Fahed, MD, MPH, Interventional Cardiologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025P001499; R01HL164629 (NIH)
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease
Keywords: Polygenic risk; Atherosclerosis; Genetics; Genomic medicine; Polygenic score; Precision medicine; Preventive cardiology; Polygenic risk score; CAD PRS
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Genetic Risk Score

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, non-inferiority trial with two parallel groups: immediate disclosure of non-high coronary artery disease polygenic risk score (CAD PRS) versus deferred disclosure after 12 months.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Disclosure (Experimental): Participants are randomized to receive their non-high CAD PRS immediately after genotyping.
  Interventions: Behavioral: Immediate disclosure of non-high CAD PRS
- Deferred Disclosure (Active Comparator): Participants are randomized to have their non-high CAD PRS withheld for 12 months before receiving their result after the follow up period.
  Interventions: Behavioral: Deferred Disclosure of non-high CAD PRS

INTERVENTIONS:
Behavioral: Immediate disclosure of non-high CAD PRS — Participants receive their non-high CAD PRS result as soon as it is available after genotyping.
  Arms: Immediate Disclosure
Behavioral: Deferred Disclosure of non-high CAD PRS — Participants receive their non-high CAD PRS result after completion of the 12 month follow up period.
  Arms: Deferred Disclosure

SUMMARY:
The goal of this clinical trial is to evaluate whether disclosure of a non-high polygenic risk score for coronary artery disease (CAD PRS) is non-inferior to standard of care in maintaining cardiovascular health over one year among adults aged 40-75 years without cardiovascular disease and not on statins.

DETAILED DESCRIPTION:
The main question PROACT 3 aims to answer is whether disclosure of a non-high CAD PRS result influences cardiovascular health behaviors and outcomes.

This is a single-center, randomized, non-inferiority trial of 400 adults aged 40-75 without cardiovascular disease and not on statins, identified through the Mass General Brigham primary care network. All participants will undergo CAD PRS testing, and those with non-high genetic risk will be randomized in a 1:1 ratio to receive immediate disclosure of their results or deferred disclosure after 12 months. The primary outcome is the change in cardiovascular health as measured by the American Heart Association's Life's Essential 8 (LE8) score from baseline to 12 months.

Secondary outcomes include engagement with preventive care, such as completion of lipid panels and blood pressure measurements, attendance at primary care visits, and initiation of preventive therapies (antihypertensive, lipid-lowering, or GLP-1 receptor agonist therapy or other anti-diabetic therapy) when clinically indicated. Additional outcomes will include changes in individual LE8 behavioral components (physical activity, diet, tobacco use, and sleep) and BMI from baseline to 12 months.

This trial is designed to address concerns about potential false reassurance from non-high CAD PRS disclosure and will provide empirical evidence to guide best practices for polygenic risk communication in preventive cardiology.

ELIGIBILITY:
Inclusion Criteria:

* Current age 40-75 years
* Established primary care at Mass General Brigham with at least one visit in the last 2 years

Exclusion Criteria:

* High CAD PRS
* Known cardiovascular disease, defined by a diagnosis of coronary artery disease, peripheral artery disease, or cerebrovascular disease
* Currently taking LDL cholesterol- lowering or anti-inflammatory medications, including statins or colchicine
* Liver disease (cirrhosis, active hepatitis, ALT > 3x ULN, total bilirubin > 2x ULN and not Gilbert's Syndrome)
* Contraindication to taking colchicine or rosuvastatin (allergy, liver or kidney disease)
* Pregnancy, breastfeeding, or planning to become pregnant during the study period
* Inability to provide informed consent
* Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m²
* BMI ≥ 40 kg/m²
* Inability to hold breath for 10 seconds

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Change in Life's Essential 8 (LE8) score from baseline to 12 months | 12 months
  The primary outcome of this study is the change in total cardiovascular health as measured by the LE8 score from baseline to 12 months. The LE8 score integrates four health behaviors (diet, physical activity, nicotine exposure, and sleep) and four health factors (body mass index, blood lipids, blood glucose, and blood pressure) into a single metric ranging from 0 (poor health) to 100 (ideal health). The trial will assess whether disclosure of a non-high CAD PRS preserves cardiovascular health within a pre-specified 5 point non-inferiority margin.

SECONDARY OUTCOMES:
Completion of lipid panel and blood pressure measurement within 12 months | 12 months
  Proportion of participants who complete a lipid panel and have blood pressure measured within 12 months of randomization, based on electronic health record data will be compared between the two groups to assess engagement with preventive care.
Attendance at primary care visit within 12 months | 12 months
  Proportion of participants attending at least one primary care visit within 12 months of randomization, as documented in the electronic health record, will be compared between the two groups to assess engagement with routine medical care.
Initiation of preventive therapies within 12 months | 12 months
  Proportion of participants initiating antihypertensive, lipid-lowering, GLP-1 receptor agonist, or other anti-diabetic therapy within 12 months when clinically indicated, based on prescription records, will be compared between the two groups to assess proactive management of cardiovascular risk factors.
Change in individual LE8 behavioral components from baseline to 12 months | 12 months
  Change in physical activity, diet, tobacco use, and sleep health from baseline to 12 months, as assessed by self-reported survey responses and calculated as individual components of the LE8 score, will be compared between the two groups to assess differences in health behaviors.
Change in body mass index (BMI) from baseline to 12 months | 12 months
  Change in BMI, calculated from height and weight measurements obtained from electronic health records, will be compared between the two groups to assess differences in weight management.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be tabulated and analyzed. Study site will not share any of the subject identifiers.